CLINICAL TRIAL: NCT03576651
Title: A Phase I, Double-blind, Randomized, Parallel-group, Single-dose, Three-Arm Study to Compare the Pharmacokinetics and to Evaluate the Tolerability, Safety and Immunogenicity of JHL1149 and Bevacizumab (Avastin) in Healthy Male Volunteers
Brief Title: A Study to Compare the Pharmacokinetics of JHL1149 and Bevacizumab (Avastin) in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: JHL Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JHL-CLIN-1149-01
Record Dates: First submitted 2018-06-25; First posted 2018-07-03 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Healthy Male Subjects
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- JHL1149 (Experimental)
  Interventions: Biological: JHL1149
- US-sourced-Avastin™ (Active Comparator)
  Interventions: Biological: Bevacizumab
- EU-sourced Avastin™ (Active Comparator)
  Interventions: Biological: Bevacizumab

INTERVENTIONS:
Biological: JHL1149 — Each patient may receive single dose of JHL1149 1mg/kg by intravenous infusion
  Arms: JHL1149
Biological: Bevacizumab — Each patient may receive single dose of Avastin 1mg/kg by intravenous infusion
  Arms: US-sourced-Avastin™
Biological: Bevacizumab — Each patient may receive single dose of Avastin 1mg/kg by intravenous infusion
  Arms: EU-sourced Avastin™

SUMMARY:
This is a Phase I, Double-blind, Randomized, Parallel-group, Single-dose, Three-Arm Study to Compare the Pharmacokinetics and to Evaluate the Tolerability, Safety and Immunogenicity of JHL1149 and Bevacizumab (Avastin) Sourced from the European Union (EU) and the Union States (US) in Healthy Male Volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteers,
2. Age range of 21-55 years (inclusive).
3. BMI range of 18.0-30.0 kg/m2 (inclusive) and a total body weight >50 kg.
4. Medically healthy subjects with normal organ functions and laboratory values
5. Subjects must be willing to use adequate contraception and not donate sperm from admission to clinical research center until 6 months post dosing.
6. All intermittent medications including over the counter, herbal and nutriceuticals, must be stopped at least 14 days prior to admission to the clinical research center.
7. Ability and willingness to abstain from alcohol 48hrs prior to admission to the clinical research center, and throughout the dosing and evaluation period.
8. No significant medical history per the PI judgment.
9. ECGs (via 12 lead) showing normalized cumulative sum (NCS) findings per PI judgment
10. Ability to provide informed consent for the study.

Exclusion Criteria:

1. Previous treatment with an anti-vascular endothelial growth factor (VEGF) antibody or any other antibody or protein targeting the VEGF receptor or treatment with an immunobiological drug during the last three months.
2. Previous history of cancer other than adequately treated basal cell or squamous cell carcinoma of the skin.
3. Received blood transfusions and blood donation within 3 months before screening date.
4. Resting blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg.
5. Any other severe physical incapacity.
6. Positive serological test for hepatitis B surface antigen or positive antibody for hepatitis C virus or positive antibody for human immunodeficiency virus (type 1 and 2).
7. Tuberculosis (TB) or an acute systemic infection; demonstrated by positive QuantiFERON-TB and/or Chest radiograph conducted up to 3 months prior or during the screening visit.
8. Major surgery planned for the study duration or cases with major surgery in the past 28 days before screening.
9. History of relevant drug and/or food related allergies.
10. History of or known hypersensitivity to bevacizumab or other recombinant human or humanized antibodies or inactive ingredients.
11. History of alcohol and or drug abuse/addiction.
12. Positive alcohol breath test and drug screen for opiates, methadone, cocaine, amphetamines, cannabinoids, barbiturates, benzodiazepines.
13. Strenuous exercise 96 hrs prior to admission to the clinical research center.
14. Any significant or acute illness within 30 days prior to the expected first dose of study drug.
15. Unsuitable veins for infusion and/or venepuncture.
16. History of bleeding disorders, thromboembolic conditions, gastrointestinal perforations or any fistulae, orthostatic hypotension, fainting spells, blackouts for any reasons; as well as presence of a non-healing wound or fracture.
17. Participation in another clinical study where the investigational drug was received within < 5 x half-lives of the drug (120 days prior to screening).
18. Any condition or displayed behaviour that the investigator in their best clinical judgement believes could be detrimental the subject's participation in the study or result in unfavourable outcomes for the subject or study (eg. Clear signs that the patient is withholding information on their substance use/abuse status).

Ages: 21 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 154 (Actual)
Dates: Start 2018-03-24 (Actual); Primary Completion 2018-09-17 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
AUC0-inf | up to 71 days
  area under the concentration-time curve from time zero to infinity (AUC0-inf)

SECONDARY OUTCOMES:
AUClast | up to 71 days
  Area under the serum concentration-time curve from time 0 to last quantifiable concentration (AUClast).
Cmax | up to 71 days
  Maximum serum concentration just prior to end of infusion (Cmax)

CONTACTS AND LOCATIONS:
Locations (1):
- MHAT Lyulin EAD, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: Undecided